CLINICAL TRIAL: NCT01724606
Title: Whole Brain Radiotherapy (WBRT) With Sorafenib for Breast Cancer Brain Metastases (BCBM): A Phase I Study
Brief Title: Whole Brain Radiotherapy (WBRT) With Sorafenib for Breast Cancer Brain Metastases (BCBM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-046
Record Dates: First submitted 2012-11-05; First posted 2012-11-12 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: Whole Brain Radiotherapy (WBRT); Sorafenib (BAY 43-9006); 12-046
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Sorafenib

ARMS (1):
- Radiotherapy with Sorafenib (Experimental): This is a single institution, open label, prospective, phase I clinical trial using standard 3+3 design. Histologically confirmed metastatic adenocarcinoma of the breast with radiologic evidence of new and/or progressive brain metastases (BM) with a clinical indication for WBRT will be enrolled.
  Interventions: Radiation: Whole Brain Radiotherapy (WBRT); Drug: Sorafenib

INTERVENTIONS:
Radiation: Whole Brain Radiotherapy (WBRT) — WBRT (30 Gy) will be delivered in 10 fractions. Standard opposed lateral fields with multileaf collimation blocking will be used. Treatment will be administered on business days and delivered over an approximate 2 week period. Dexamethasone may be given at the discretion of the treating physician but the dose cannot exceed greater than 16mg daily as it is a strong CYP3A4 inducer. Patients will also receive a proton pump inhibitor with dexamethasone.
Drug: Sorafenib — The proposed three dose levels of sorafenib during dose escalation are 200 mg, 400mg, and 600 mg administered daily orally. Patients will be enrolled in cohorts of 3.The first three subjects will take sorafenib 200 mg daily within a few hours after the first RT fraction. Sorafenib will be continued concurrently with WBRT (1 fraction /day x 10 fractions) without breaks and then continued after WBRTfor a total of 21 days. If no dose limiting toxicity (DLT) is observed in a cohort of 3 patients until two weeks after completion of WBRT, the next dose level will be evaluated.

SUMMARY:
Sorafenib is a new type of anti-cancer drug. It belongs to a new class of medications known as tyrosine kinase inhibitors. Sorafenib is thought to work against cancer in many ways. It helps decrease blood supply to the tumor. It also blocks some proteins that help the tumor cells to grow." Sorafenib is approved by the Food and Drug administration (FDA) for treatment for other cancers like liver and kidney cancer. Sorafenib has also been studied in the treatment of breast cancer that has spread but is not specifically approved for the treatment of breast cancer. It has been studied both as a single agent and also in combination with other anti-cancer therapies for breast cancer. In laboratory models and in some patients with other cancers, sorafenib has been studied in tumors in the brain.

In this study, sorafenib will be given together with whole brain radiation therapy (WBRT). Overall this research study is designed to answer 2 main questions:

1. What dose of sorafenib should be used together with WBRT?
2. What are the side effects of sorafenib and WBRT when given together?

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed metastatic adenocarcinoma of the breast (Confirmation will be done at MSKCC)
* Age ≥18 years.
* Radiologic evidence of new and/or progressive brain metastasis (≥10 mm in longest dimension) by MR imaging of the Brain
* Life expectancy of >12 weeks.
* Karnofsky Performance Status (KPS) of ≥70%
* If a patient is on corticosteroids, he/she must be on a non-escalating corticosteroid dose (not exceeding more than 16 mg daily of Dexamethasone oral) for ≥ 5 days.
* No limit to prior therapies with last anti-cancer treatment ≥ 2 weeks from initiation of protocol based therapy provided all toxicities (other than alopecia) have resolved to ≤Grade 1 or baseline.
* Planned WBRT based on number (≥ 3 lesions) and/or size (≥ 1 cm) of BMs (SRS) in addition to WBRT will also be eligible.
* Patients with prior SRS will also be eligible, provided that there are new, non-irradiated measurable brain lesions.
* No limit to prior therapies with last anti-cancer treatment ≥2 weeks from initiation of WBRT. Please note: there is no washout period required for trastuzumab and pertuzumab.
* Prior hormonal therapy for locally advanced or metastatic disease is allowed but this must have been discontinued prior to enrollment. No washout period will be required.
* Continuation of trastuzumab and pertuzumab are allowed for those patients already on trastuzumab and pertuzumab therapy.
* Adequate bone marrow, liver, and renal function as assessed by the following:
* Granulocyte count ≥ 1,000/μL, platelet count ≥ 100,000/μL, and hemoglobin ≥ 10 g/dL (hematologic parameters must be assessed at least 14 days after a prior transfusion, if any)
* Serum bilirubin ≤ 1.5 mg/dL; AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN except for: Patients with hepatic metastases: ALT and AST ≤ 5 × ULN; patients with hepatic and/or bone metastases:
* alkaline phosphatase ≤ 5 × ULN and patients with Gilbert's disease: serum bilirubin < 5 mg/dL
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance of ≥ 60 mL/min based on a 24-hour urine collection
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to enrollment and must agree to use adequate contraception prior to enrollment and for the duration of study participation. Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug.
* Patients must be able to swallow and retain oral medication.

Exclusion Criteria:

* Leptomeningeal metastases, hemorrhagic metastases, presence of midline shift Please note: leptomeningeal metastases may be allowed if it is limited to cranial metastasis (MRI spine should be completed, within 4 weeks of enrollment, to show that no other leptomeningeal metastases is present) and is not the only metastasis present in the brain.'
* Contraindications to sorafenib
* Prior treatment with any agent that targets vascular endothelial growth factor (VEGF) or VEGF receptors (VEGFR) (licensed or investigational including sorafenib), except bevacizumab.
* Craniotomy or any other major surgery, open biopsy, or significant traumatic injury within 4 weeks of enrollment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Uncontrolled seizures
* Use of cytochrome P450 enzyme-inducing anti-epileptic drugs (such as phenytoin, carbamazepine, or phenobarbital) is not allowed.
* Cardiac disease:
* Congestive heart failure >class II New York Heart Association (NYHA) (See Appendix B, or
* Unstable angina (anginal symptoms at rest), or new-onset angina (begun within the last 3 months), or myocardial infarction within the 6 months prior to enrollment, or
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Congenital long QT syndrome or taking drugs known to prolong the QT interval ( See Appendix D or http://www. Azcert.org )
* Subjects taking any drugs with a known risk of causing torsades de pointes.
* Grade 3 hypertension ( SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg despite maximal medical therapy)
* ≥ Grade 2 Lipase increased (>1.5 x ULN),
* Thrombolic, embolic, venous, or arterial events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Evidence or history of bleeding diathesis or coagulopathy at the time of enrollment.
* Pulmonary hemorrhage/bleeding event >National Cancer Institute Common Terminology for Adverse Events (NCI-CTCAE, version 4.0) Grade 2 within 4 weeks of enrollment.
* Any other hemorrhage/bleeding event ≥NCI-CTCAE Grade 3 within 4 weeks of enrollment.
* Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin) or with heparins and heparinoids. However, prophylactic anticoagulation as described below is allowed:
* Low dose warfarin (1 mg orally, once daily) with PT-INR ≤ 1.5 x ULN is permitted. Infrequent bleeding or elevations in PT-INR have been reported in some subjects taking warfarin while on sorafenib or capecitabine therapy. Therefore, subjects taking concomitant warfarin should be monitored regularly for changes in PT, PT-INR or clinical bleeding episodes.
* Low dose aspirin (≤ 100 mg daily).
* Active clinically serious infection >NCI-CTCAE Grade 2.
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C (the safety and effectiveness of sorafenib in this patient population have not been studied).
* Previous or concurrent cancer that is distinct in primary site or histology from breast cancer within 5 years prior to enrollment EXCEPT cervical cancer in situ, treated basal cell carcinoma, squamous cell carcinoma (SCC), as long as it is other than SCC involving skin of the head and/or neck, and superficial bladder tumors [Ta and Tis].
* Subjects who have used strong CYP3A4 inducers (eg, phenytoin, carbamazepine, phenobarbital, St. John's Wort [Hypericum perforatum], dexamethasone at a dose of greater than 16 mg daily for more than one day, or rifampin [rifampicin], and/or rifabutin) within 28 days before randomization.
* Concurrent anti-cancer therapy (chemotherapy, hormonal therapy, radiation therapy (other than that specified by the protocol), surgery, immunotherapy, biologic therapy including trastuzumab, lapatinib, bevacizumab, tyrosine kinase inhibitors other than sorafenib or tumor embolization
* Women who are pregnant or breast-feeding.
* Use of any investigational drug within 28 days or 5 half-lives, whichever is longer, preceding enrollment. For the purposes of this study, bevacizumab will not be considered investigational therapy.
* Inability to comply with protocol and /or not willing or not available for follow-up assessments.
* Any condition which in the investigator's opinion makes the patient unsuitable for the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 year
  Dose-escalation Phase: The proposed three dose levels of sorafenib during dose escalation are 200 mg, 400mg, and 600 mg administered daily orally. The dose-escalation phase is for 3-6 patients to be treated at each dose level. Assuming 3 dose levels during this phase, it will require a minimum of 2 and a maximum of 18 patients.
assessing toxicity by the number of adverse events | 1 year
  using the active version of the CTCAE version 4.0

SECONDARY OUTCOMES:
CNS progression-free survival | 1 year
  CNS-PFS is defined as the interval between the date of study entry and the date of intracranial tumor progression or death from any cause. We will evaluate this during follow-up MRI scans that will be performed as a standard of care using the Macdonald criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/